CLINICAL TRIAL: NCT02103829
Title: "Quit Smoking on Your Own" Brief Online Study
Acronym: TC-PAU-1
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: i4Health (Other)
Responsible Party: Principal Investigator, Ricardo F. Muñoz, Ph.D., Distinguished Professor of Clinical Psychology, i4Health
Allocation: Randomized | Model: Factorial | Masking: None
Other Study IDs: TC-PAU-1
Record Dates: First submitted 2014-04-01; First posted 2014-04-04 (Estimated); Last update posted 2016-09-29 (Estimated); Status verified 2016-09

CONDITIONS: Cigarette Smoking
Keywords: Cigarette smoking; Tobacco smoking; Smoking, Tobacco
MeSH Terms: conditions — Cigarette Smoking; Tobacco Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Condition #1 (Active Comparator): Condition #1 will consist of Brief Intervention #1, a brief online suggestion that takes less than 1 minute to complete.
  Interventions: Behavioral: Brief Intervention #1
- Condition #2 (Experimental): Condition #2 will consist of Brief Intervention #1 and Brief Intervention #2 that together take less than a minute to complete.
  Interventions: Behavioral: Brief Intervention #1; Behavioral: Brief Intervention #2
- Condition #3 (Experimental): Condition #3 will consist of Brief Intervention #1 and Brief Intervention #3, which, together, will take less than 8 minutes to complete.
  Interventions: Behavioral: Brief Intervention #1; Behavioral: Brief Intervention #3
- Condition #4 (Experimental): Condition #4 will consist of Brief Intervention #1, Brief Intervention #2, and Brief Intervention #3, which, together, will take less than 8 minutes to complete.
  Interventions: Behavioral: Brief Intervention #1; Behavioral: Brief Intervention #2; Behavioral: Brief Intervention #3

INTERVENTIONS:
Behavioral: Brief Intervention #1 — Brief online suggestion intended to increase the likelihood of quitting smoking that takes less than 1 minute to complete.
Behavioral: Brief Intervention #2 — Brief online suggestion intended to increase the likelihood of quitting smoking that takes less than 1 minute to complete.
  Arms: Condition #2; Condition #4
Behavioral: Brief Intervention #3 — Brief online suggestion intended to increase the likelihood of quitting smoking that takes less than 7 minutes to complete.
  Arms: Condition #3; Condition #4

SUMMARY:
Most individuals who smoke want to quit smoking. Most individuals who want to quit, quit on their own. The purpose of this study is to determine whether very brief suggestions provided online are comparatively more effective than others in increasing motivation to quit immediately after the suggestions are implemented and actual quit rates one month later.

There are no costs associated with participating in this study and participants will not be compensated for their participation.

To join the study paste the following link into your browser:

https://www.i4health-pau.org/quit-smoking-on-your-own

The entire study takes place online on an automated website.

DETAILED DESCRIPTION:
Participants will be recruited online using search engine ads (e.g., Google), online association list serves, community websites designed to reach individuals interested in participating in research studies, and social media sites related to smoking cessation efforts.

The entire study will be administered online. Participants may complete it at a time and place of their convenience.

To join the study paste the following link into your browser:

https://www.i4health-pau.org/quit-smoking-on-your-own

The website will automatically obtain consent, ask 16 brief questions as a pre-test, randomize to 4 very brief interventions, ask 4 post-test questions, and at 1-month follow-up, send an email with a link to a 6-question survey. The initial online session is expected to take between 3 and 8 minutes and the 1-month follow-up survey less than 2 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Adult (18 years of age or older)
* Smoker who wants to quit
* Access to the Internet

Exclusion Criteria:

* Less than 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 345 (Actual)
Dates: Start 2014-03; Primary Completion 2016-02 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Percentage of participants who report quitting smoking | 1 month
  Percentage of respondents who respond "no" to the question: "Have you smoked 1 or more cigarettes in the last 7 days?"

SECONDARY OUTCOMES:
Motivation to quit smoking | 10 minutes
  Pre-post measure of motivation before and after the brief suggestions being tested are administered online. Specifically, response on a 0 to 10 scale (from "not at all" to "extremely") to the question "How motivated are you to stop smoking in the next 4 weeks?"

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo F Muñoz, Ph.D., Principal Investigator — Palo Alto University
Locations (1):
- Palo Alto University i4Health, Palo Alto, California, United States